CLINICAL TRIAL: NCT06179108
Title: A Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Evaluate the Antipsychotic Efficacy and Safety of LB-102 in the Treatment of Adult Patients With Acute Schizophrenia
Brief Title: Randomized, Double-blinded, Placebo-controlled, Evaluating the Treatment With LB-102 in Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LB Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB-102-003
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 3:3:3:1 to receive with placebo (n ~ 105), 50 mg LB-102 QD (n ~ 105), 75 mg LB-102 QD (n ~ 105), 100 mg LB-102 QD (n ~ 35) orally.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LB-102, 50 mg QD (Experimental): Oral LB-102: 50 mg (n ~ 105)
  Interventions: Drug: LB-102
- LB-102, 75 mg QD (Experimental): Oral LB-102: 75 mg (n ~ 105)
  Interventions: Drug: LB-102
- LB-102, 100 mg (Experimental): Oral LB-102: 100 mg (n ~ 35)
  Interventions: Drug: LB-102
- Placebo comparator (Placebo Comparator): Drug: Placebo
  Matched placebo tablets
  Interventions: Drug: LB-102

INTERVENTIONS:
Drug: LB-102 — LB-102 is a dopamine D2/3 and 5HT7 antagonist.

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multi-center inpatient study to evaluate the efficacy and safety of LB-102 in adult patients diagnosed with acutely exacerbated schizophrenia. To determine whether LB-102 administered to patients with acutely exacerbated schizophrenia demonstrates antipsychotic efficacy, as determined by a change from Baseline on the Positive and Negative Syndrome Scale (PANSS) total score, compared to placebo at 28 days. The secondary objectives of the study are to evaluate improvement in CGI-S, safety and tolerability, and pharmacokinetics.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multi-center inpatient study to examine the efficacy and safety of LB-102 in adult patients diagnosed with acutely exacerbated schizophrenia. The primary objective of the study is to assess the efficacy of LB-102 versus placebo in reducing Positive and Negative Syndrome Scale (PANSS) total scores at day 28 in approximately 350 adult inpatients with a DSM-5 diagnosis of schizophrenia. The secondary objectives of the study are to evaluate improvement in CGI-S, PANSS subscale and Marder Factor scores, safety and tolerability, and pharmacokinetics in adult inpatients with a DSM-5 diagnosis of schizophrenia. The duration of treatment of the study is 28 days (4 weeks). Patients in this study will be randomized 3:3:3:1 to receive either: placebo, 50 mg QD LB-102, 75 mg QD LB-102, or 100 mg QD LB-102; that is, ~105 patients will get placebo, ~105 will get 50 mg LB-102 QD, ~105 will get 75 mg LB-102 QD, ~35 will get 100 mg LB-102 QD. LB-102 will be dosed orally once a day. Pharmacokinetic data will be measured for the first 60 patients in this study.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in the study if they meet all of the following criteria:

1. Patient who is able to provide written informed consent (as required by Institutional Review Board [IRB]) prior to the initiation of any protocol-required procedures.
2. Must be willing to be hospitalized for the duration of the inpatient period of the study.
3. Have stable living environment when not in a hospital.
4. Male and female patients 18 to 55 years of age inclusive at the time of informed consent with a diagnosis of schizophrenia as defined by DSM-5 criteria and confirmed by the MINI 7.0.2 .
5. Body mass index (BMI) must be ≥18 and ≤40 kg/m2.
6. Patient who experiencing an acute exacerbation of psychotic symptoms, AND the patient requires hospitalization OR if already an inpatient at Screening, has been hospitalized for onset < 2 weeks for the current exacerbation.
7. Patients who are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by meeting ALL of the following criteria at the Screening and Baseline visits:

   * Total PANSS score between 80 and 120, inclusive, and
   * Score of ≥4 (moderate or greater) for ≥2 of the following Positive Scale (P) items: Item 1 (P1; delusions), Item 2 (P2; conceptual disorganization), Item 3 (P3; hallucinatory behavior), Item 6 (P6; suspiciousness/persecution), and
   * CGI-S score ≥4 (moderately to severely ill).
8. Have received previous antipsychotic treatment (dose and duration as per the label) and who showed a previous good response to such antipsychotic treatment (other than clozapine) in the last 12 months, according to the Investigator's opinion.
9. Have history of relapse and/or exacerbation of symptoms when they were not receiving antipsychotic treatment.
10. Patients willing to discontinue all prohibited psychotropic medications prior to Screening, if determined to be clinically appropriate by the Investigator, and not for the sole purpose of inclusion in the trial.

Exclusion Criteria:

A patient will be excluded from the study if they meet any of the following criteria:

Sex and Reproductive Status

1. Sexually active females of childbearing potential and male patients who are not practicing 2 different methods of birth control with their partner during the trial and for 30 days after the last dose of trial medication or who would not remain abstinent during the trial and for 30 days after the last dose.
2. Females who are breastfeeding or who have a positive pregnancy test result prior to receiving trial medication.
3. Patients who presented with a first episode of schizophrenia.
4. Improvement of ≥20% in total PANSS score between the Screening and Baseline assessments.
5. History of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (dose and duration as per the label) or required clozapine within the last 12 months.
6. Current DSM-5 Axis I diagnosis other than schizophrenia.
7. Risk for suicidal behavior during the study.
8. Risk of violent or destructive behavior.
9. Patients with clinically significant tardive dyskinesia.
10. Patients with a score of 3 on the Barnes Akathisia Rating Scale (BARS) global clinical assessment of akathisia.
11. Patients who met DSM-5 criteria for substance abuse or dependence within the past 1 year.
12. Patients with hypothyroidism or hyperthyroidism or clinically significant abnormal thyroid function.
13. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
14. Patients with insulin-dependent diabetes mellitus (i.e., any patient using insulin) are excluded. Patients with non-insulin-dependent diabetes mellitus may be eligible for the trial if their condition is stable as determined by satisfying ALL of the following criteria:

    * Glycosylated hemoglobin (HbA1c) <7.0%, and
    * Screening glucose must have been ≤125 mg/dL or ≤6.94 mmol/L (fasting) or <200 mg/dL or <11.1 mmol/L (nonfasting), and
    * Patient had been maintained on a stable regimen of oral antidiabetic medication(s) for at least 28 days prior to Screening or diabetes had been well controlled by diet for at least 28 days prior to Screening, and
    * Patient had no hospitalizations within the 12 months prior to Screening due to diabetes or complications related to diabetes, and
    * Patient's diabetes should not be newly diagnosed during Screening for the trial.
15. Patients with uncontrolled hypertension or symptomatic hypotension, or orthostatic hypotension
16. Patients with known ischemic heart disease or any history of myocardial infarction, congestive heart failure.
17. Patients with epilepsy or a history of seizures.
18. Patients with a positive urine drug screen or a positive blood alcohol test.
19. Patients with a history of alcohol use or substance use disorder (by DSM-5 criteria) within 12 months of Screening or a positive screen for drugs of abuse at Screening.
20. The following laboratory test results are exclusionary:

    * Platelets ≤75,000/µL or ≤75×109/L
    * Hemoglobin ≤9 g/dL or ≤90 g/L
    * Neutrophils, absolute ≤1000/µL or ≤1×109/L
    * AST and ALT >2 × upper limit of normal (ULN)
    * CPK >3 × ULN, unless discussed with and approved by the Medical Monitor
    * Creatinine ≥2 mg/dL or ≥176.8 µmol/L
    * Estimated creatinine clearance of <45 mL/min, calculated using the Cockcroft-Gault equation, at Screening
    * HbA1c ≥7.0%
    * Abnormal free T4 (during Screening), unless discussed with and approved by the Medical Monitor.
21. Clinically significant abnormal finding on the triplicate set of electrocardiograms (ECGs) or evidence of any of the following cardiac conduction abnormalities at Screening.
22. Patients who are currently taking oral antipsychotic medications, monoamine oxidase inhibitors (MAOIs), anticonvulsants (e.g., lamotrigine, Depakote), tricyclic antidepressants (e.g., imipramine, desipramine), selective serotonin reuptake inhibitors, and any other antidepressants or any other psychoactive medications (except lorazepam, zolpidem, zaleplon, eszopiclone, or similar benzodiazepines, diphenhydramine, benztropine, and propranolol). The medications should not be discontinued solely to make the patient eligible for enrollment in the study.
23. Patients who received electroconvulsive therapy, or Transcranial Magnetic Stimulation (TMS).
24. Patients with a history of neuroleptic malignant syndrome.
25. Patients with a history of allergic response
26. Prisoners or patients who were compulsorily detained (involuntarily hospitalized) for treatment of either a psychiatric or physical illness or have been in the last 6 months prior to the Screening Visit
27. Patients who have participated in another clinical study in which they received an experimental or investigational drug agent within 3 months of Screening.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 359 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (25):
- United States (25):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodland Internation Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - CelExel Clinical Innovations, Bellflower, California
  - Synexus, Cerritos, California
  - ProScience Research Group, Culver City, California
  - CelExel CNS, Garden Grove, California
  - Synergy Research, Lemon Grove, California
  - CenExel CIT Riverside, Riverside, California
  - NRC Research Institute, Santa Ana, California
  - Behavioral Clinical Research, Inc., Hollywood, Florida
  - CenExel RCA, Hollywood, Florida
  - Segal Institute for Clinical Research, Miami Lakes, Florida
  - CenExel ACMR, Atlanta, Georgia
  - CenExel iResearch, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Pillar Clinical Research, Chicago, Illinois
  - CenExel CBH, Gaithersburg, Maryland
  - CenExel HRI, Berlin, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Community Clinical Research, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Pillar Clinical Research, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grattan V, Vaino AR, Prensky Z, Hixon MS. Antipsychotic Benzamides Amisulpride and LB-102 Display Polypharmacy as Racemates, S Enantiomers Engage Receptors D2 and D3, while R Enantiomers Engage 5-HT7. ACS Omega. 2019 Aug 15;4(9):14151-14154. doi: 10.1021/acsomega.9b02144. eCollection 2019 Aug 27. PMID 31497735
- [Background] Biernat L, Grattan VT, Hixon MS, Prensky Z, Vaino AR. A randomized, double-blind, placebo controlled, phase 1 study of the safety, tolerability, pharmacokinetics, and pharmacodynamics of LB-102, a selective dopamine D2/3/5-HT7 inhibitor. Psychopharmacology (Berl). 2022 Sep;239(9):3009-3018. doi: 10.1007/s00213-022-06185-7. Epub 2022 Jul 16. PMID 35841422

RESULTS

PARTICIPANT FLOW:
Groups:
- LB-102, 50 mg QD: Oral LB-102: 50 mg (n = 107)
- LB-102, 75 mg QD: Oral LB-102: 75 mg (n = 108)
- LB-102, 100 mg QD: Oral LB-102: 100 mg (n = 36)
- Placebo Comparator: Matched placebo tablets (n = 108)
Period: Overall Study
Arm/Group | LB-102, 50 mg QD | LB-102, 75 mg QD | LB-102, 100 mg QD | Placebo Comparator
Started | 107 | 108 | 36 | 108
Completed | 76 | 80 | 22 | 83
Not Completed | 31 | 28 | 14 | 25
Not completed — Withdrawal by Subject | 16 | 19 | 10 | 11
Not completed — Lost to Follow-up | 12 | 4 | 1 | 9
Not completed — Adverse Event | 2 | 3 | 3 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- LB-102, 50 mg QD; LB-102, 75 mg QD; LB-102, 100 mg; Placebo Comparator: 1 tablet daily for 28 days
- Total: Total of all reporting groups
Arm/Group | LB-102, 50 mg QD | LB-102, 75 mg QD | LB-102, 100 mg | Placebo Comparator | Total
Number analyzed (Participants) | 107 | 108 | 36 | 108 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.64) | 39.2 (9.17) | 39.1 (9.19) | 39.1 (9.11) | 39.1 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 8 | 23 | 69
  Male | 87 | 90 | 28 | 85 | 290
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 87 | 83 | 25 | 80 | 275
  White | 17 | 18 | 9 | 24 | 68
  More than one race | 2 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 1 | 2 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in the PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a scale used for measuring symptom severity of patients with schizophrenia. The PANSS rating is composed of 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Patients are scored from 1 to 7 on each symptom scale. The total score of the PANSS is a minimum of 30 and a maximum of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms whereas a higher PANSS total value represents a worse outcome
Time Frame: Baseline to Day 28 (4 weeks)
Population: N for analyzed participants reflects all participants (i.e., including those with missing data imputed). Missing PANNS total scores were imputed using a mixture of MAR and MNAR approaches depending on the reason for missingness.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- LB-102, 100 mg: Oral LB-102: 100 mg (n = 36)
Arm/Group | LB-102, 50 mg QD | LB-102, 75 mg QD | LB-102, 100 mg | Placebo Comparator
Number analyzed (Participants) | 107 | 108 | 36 | 108
score on a scale | -14.28 (1.097) | -13.95 (1.108) | -16.08 (1.906) | -9.27 (1.078)
Statistical Analysis 1: Comparison: LB-102, 50 mg QD vs Placebo Comparator; Test type: Superiority; p = 0.0009, Mixed Models Analysis — Hochberg's step-down procedure was adopted to control type I error across the 50 and 75 mg arms; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline total PANSS score
Statistical Analysis 2: Comparison: LB-102, 75 mg QD vs Placebo Comparator; Test type: Superiority; p = 0.0022, Mixed Models Analysis — Hochberg's step-down procedure was adopted to control type I error across the 50 and 75 mg arms; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline total PANSS score
Statistical Analysis 3: Comparison: LB-102, 100 mg vs Placebo Comparator; Test type: Superiority; p = .0017, Mixed Models Analysis; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline total PANSS score

2. Secondary Outcome: Change From Baseline to Week 4 in the CGI-S Score
Description: The Clinical Global Impressions-Severity (CGI-S) rates illness severity on a scale from 1 to 7 and has been shown to correlate with PANSS.
  The CGI-S is rated on a 7-point scale commonly used in clinical settings and research to evaluate the severity of symptoms and treatment responses in patients with mental disorders. The CGI-S specifically focuses on the severity of illness at the time of assessment, where clinicians assess the patient's current condition relative to their past. The scoring is for the CGI-S:1-normal, not at all ill, 2-Borderline mentally ill, 3-Mildly ill, 4-Moderately ill, 5-Markedly ill, 6-Severely ill, and 7-Extremely ill. The higher the score the more ill the patient is.
Time Frame: 28 days
Population: N for Analyzed participants reflects observed CGI-S data at Week 4.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LB-102, 50 mg QD | LB-102, 75 mg QD | LB-102, 100 mg | Placebo Comparator
Number analyzed (Participants) | 91 | 83 | 23 | 94
score on a scale | -.72 (0.076) | -.67 (0.075) | -.84 (0.136) | -.39 (0.074)
Statistical Analysis 1: Comparison: LB-102, 50 mg QD vs Placebo Comparator; Test type: Superiority; p = 0.0008, Mixed Models Analysis; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline CGI-S score
Statistical Analysis 2: Comparison: LB-102, 75 mg QD vs Placebo Comparator; Test type: Superiority; p = 0.0048, Mixed Models Analysis; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline CGI-S score
Statistical Analysis 3: Comparison: LB-102, 100 mg vs Placebo Comparator; Test type: Superiority; p = 0.0026, Mixed Models Analysis; MMRM included treatment group, pooled study site, visit, visit by treatment interaction and baseline CGI-S score

ADVERSE EVENTS:
Time Frame: From Screening to study day 56
Arm/Group | LB-102, 50 mg QD | LB-102, 75 mg QD | LB-102, 100 mg QD | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/108 | 0/36 | 1/108
Serious Adverse Events (participants affected / at risk) | 1/107 | 1/108 | 1/36 | 2/108
Other Adverse Events (participants affected / at risk) | 74/107 | 62/108 | 27/36 | 60/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LB-102, 50 mg QD (N=107) | LB-102, 75 mg QD (N=108) | LB-102, 100 mg QD (N=36) | Placebo Comparator (N=108)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Exacerbation of psychosis
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LB-102, 50 mg QD (N=107) | LB-102, 75 mg QD (N=108) | LB-102, 100 mg QD (N=36) | Placebo Comparator (N=108)
Hyperprolactinaemia (Endocrine disorders) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Blood prolactin increased (Investigations) | 7 (7) | 6 (6) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 27 (37) | 23 (27) | 14 (14) | 24 (31)
Headache (Nervous system disorders) | 12 (14) | 9 (10) | 2 (2) | 10 (11)
Anxiety (Psychiatric disorders) | 10 (12) | 9 (10) | 4 (4) | 9 (10)
Agitation (Psychiatric disorders) | 11 (50) | 6 (19) | 4 (4) | 10 (29)
Weight increased (Investigations) | 13 (13) | 8 (8) | 3 (3) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT06179108/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT06179108/SAP_001.pdf